CLINICAL TRIAL: NCT04376853
Title: CoronaWatch - Early Detection of Cardiovascular Risks in COVID-19 Via SmartWatch
Acronym: CoronaWatch
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: The German Heart Foundation (Other); Klaus Tschira Stiftung, Germany (Unknown); Freunde und Förderer der Kardiologie Heidelberg; Germany (Unknown)
Responsible Party: Principal Investigator, Benjamin Meder, Prof. Dr. med., University Hospital Heidelberg
Other Study IDs: CoronaWatch
Record Dates: First submitted 2020-04-20; First posted 2020-05-06 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: COVID-19; Wearable; SmartWatch; Prognostics; Diagnostics; Risk stratification; Apple Watch
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Patients with COVID-19, who have cardiovascular diseases or receive medication with arrhythmogenic risk.
  Interventions: Device: Apple Watch Series 5

INTERVENTIONS:
Device: Apple Watch Series 5 — Digital monitoring via Apple Watch

SUMMARY:
In December 2019, a new viral disease called COVID-19 emerged. It is caused by the new corona virus SARS-CoV-2. It was initially described in the chinese city of Wuhan. In the following months, the disease developed into a pandemic, which is currently an immense international challenge.

So far, there is little scientific evidence on risk stratification, especially on the prognostic value of biomarkers (laboratory-chemical, clinical and digital) with regard to clinical deterioration of patients with COVID-19. Further scientific studies are needed to establish optimal risk stratification and early detection of clinical deterioration.

In this study, the investigators aim to observe patients with COVID-19 via SmartWatches on top of their clinical routine. The investigators aim to determine, whether the addition of SmartWatches enhances risk stratification, early detection of complications and prognostics in patients with COVID-19, who have cardiovascular diseases or receive medication with arrhythmogenic risk.

DETAILED DESCRIPTION:
In December 2019, a new viral disease called COVID-19 emerged. It is caused by the new corona virus SARS-CoV-2. It was initially described in the chinese city of Wuhan. In the following months, the disease developed into a pandemic, which is currently an immense international challenge.

So far, there is little scientific evidence on risk stratification, especially on the prognostic value of biomarkers (laboratory-chemical, clinical and digital) with regard to clinical deterioration of patients with COVID-19. Further scientific studies are needed to establish optimal risk stratification and early detection of clinical deterioration.

In this study, the investigators aim to observe patients with COVID-19 via SmartWatches on top of their clinical routine. The investigators aim to determine, whether the addition of SmartWatches enhances risk stratification, early detection of complications and prognostics in patients with COVID-19, who have cardiovascular diseases or receive medication with arrhythmogenic risk.

The study is a monocentric observational study in the sense of a cohort study. 50 COVID-19 patients are aimed to be included. Patients are identified upon presentation at the COVID-19 outpatient clinic or during their stay at the COVID-19 ward at the Centre for Internal Medicine (Krehl-Klinik) at the Heidelberg University Hospital.

Since many study-relevant data are routinely collected at presentation in the outpatient clinic or during the inpatient stay, these values are being accessed (e.g. anamnesis, physical examination, ECGs, CT and laboratory values) by our study team.

The recruited subjects (n=50) receive medical care according to the instructions of the treating physicians. The treating physicians decide whether a home or inpatient quarantine is necessary and whether a specific therapy is required.

SmartWatches are provided to all subjects on the day of recruitment. These are Apple Watches (Series 5). The patient is asked to record an ECG on the Apple Watch 5 times a day (8:00 am, 11:00 am, 2:00 pm, 5:00 pm, 8:00 pm). Furthermore, the activity of the patient is recorded via the App Health.

The data collected by the Apple Watch (activity and health-related data of the App Health as well as ECGs) are accessible to the study team at any time, provided that the pseudonymised data transfer via Email has been successfully completed. In order to be able to use the Apple Watch, participants are provided with an iPhone by us.

As soon as the COVID-19 disease is cured or the participant died, the study ends for them. However, the study will be conducted for at least 14 days for each patient, even if the patient has healed earlier.

If findings relevant to the health of the patients should arise from the study-relevant data (for example the detection of cardiac arrhythmias via the Apple Watch), the investigators report these information to the treating physician and patient as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 (detection by PCR)
* Age ≥ 18
* The patient has understood the study design and the informed consent form and has signed and dated the informed consent form
* The patient has got a cardiovascular disease or therapy with potential cardiovascular complications

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with COVID-19. The patients have got a cardiovascular disease or therapy with potential cardiovascular complications.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Biomarker | 3 months
  Identification of biomarkers (laboratory-chemical, clinical, digital) for risk stratification, early detection of complications and prognosis

SECONDARY OUTCOMES:
Protective factors | 3 months
  Identification of laboratory-chemical, clinical or digitally measured protective factors, that indicate good prognosis
SmartWatch compliance | 3 months
  The amount of time is compared between participants regarding the wearing of a SmartWatch as a monitoring tool
Arrhythmias | 3 months
  Detection of an irregular heartbeat (PPG) as a sign of atrial or ventricular arrhythmias and correlation to intermittently recorded ECGs by SmartWatch
QT time changes | 3 months
  Detection of QT time changes (prolongation) in intermittently recorded ECGs by SmartWatch and correlation with clinical variables (change of medication, fever, etc.)
Longitudinal risk models | 3 months
  Application of artificial intelligence and machine learning techniques for longitudinal risk models by using collected data (e.g. metabolomics)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Meder, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Department III of Internal Medicine, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided